CLINICAL TRIAL: NCT04066010
Title: Optimizing the Approach of Mobile Application Use to Improve Medication Adherence in Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercer University (Other)
Collaborators: Emory Healthcare (Other); Grady Health System (Other); Atlanta Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H1605145
Record Dates: First submitted 2019-08-21; First posted 2019-08-22 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Medication Adherence; Hypertension
MeSH Terms: conditions — Medication Adherence; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Other): Mobile application intervention
  Interventions: Other: Mobile application (BP-n-Me)

INTERVENTIONS:
Other: Mobile application (BP-n-Me) — The mobile app consisted of a series of features including (1) calendar reminders of when to take medications and the patient's antihypertensive medication regimen (2) a "Call your Pharmacist" button specific to patient's pharmacy, (3) a BP log in which the patient could enter blood pressure values that were automatically compared to goal values, (4) counseling points for lifestyle and adherence factors individually tailored to each patient and (5) lifestyle and medication adherence surveys.
  Arms: Intervention

SUMMARY:
The purpose of this study was to determine the effectiveness of using a custom-designed mobile application to improve blood pressure (BP) and promote adherence to antihypertensive medication regimens. This was a prospective, multicenter, randomized controlled trial. Patients were randomized to an intervention or control group for three months. Antihypertensive medication refill history was assessed three months before, during and three months after the study period. Continuous outcome measures investigated were systolic/diastolic BP and medication refill history, using the cumulative medication gap (CMG) score.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Diagnosed with hypertension as evidenced by diagnosis codes or chart documentation
* Prescribed at least one antihypertensive for a minimum of three months prior to enrollment
* Have access to an Android mobile device with data capabilities
* Consent to using the application on their device

Exclusion Criteria:

* Do not read or speak English
* Unable to read and sign the informed consent or Health Insurance Privacy and Accountability Act (HIPAA) waiver
* Too ill or cognitively impaired to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 6 months
  This was assessed based on cumulative medication gap (CMG)
Blood pressure | 6 months
  This was assessed by measuring the change of systolic and diastolic blood pressure

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555